CLINICAL TRIAL: NCT04562532
Title: Multicenter Randomized Assessment of the Firehawk™ Rapamycin TARGET Eluting Cobalt Chromium Coronary Stent System - North American Trial
Brief Title: Firehawk Rapamycin Target Eluting Coronary Stent North American Trial
Acronym: TARGET-IV_NA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGET-IV_NA
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Firehawk group (Experimental): Participants implant Firehawk stent(s)
  Interventions: Device: Microport Firehawk stent
- 2nd generation DES (Active Comparator): Participants implant Everolimus eluting stents (Xience family - Abbott Vascular, Promus family- Boston Scientific, Synergy - Boston Scientific), or Zotarolimus eluting stents (Resolute/Onyx family and Endeavor- Medtronic), or Sirolimus eluting stents (Orsiro- Biotronik)
  Interventions: Device: 2nd generation DES (XIENCE family, Promus family, Resolute/Onyx family/Endeavor, and Orsiro stent)

INTERVENTIONS:
Device: Microport Firehawk stent — MicroPort Firehawk biodegradable polymer rapamycin target eluting stent
  Other Names: MicroPort Firehawk rapamycin target eluting stent
  Arms: Firehawk group
Device: 2nd generation DES (XIENCE family, Promus family, Resolute/Onyx family/Endeavor, and Orsiro stent) — * Everolimus eluting stents (Xience family - Abbott Vascular, Promus family- Boston Scientific, Synergy - Boston Scientific)
  * Zotarolimus eluting stents (Resolute/Onyx family and Endeavor- Medtronic)
  * Sirolimus eluting stents (Orsiro- Biotronik)
  Arms: 2nd generation DES

SUMMARY:
The aim of the TARGET-IV NA trial is to demonstrate the clinical non-inferiority of the Firehawk® rapamycin eluting stent system in comparison to currently approved 2nd generation DES for the treatment of subjects with ischemic heart disease (NSTEMI, recent STEMI (>24 hours from initial presentation and in whom enzyme levels have peaked), unstable angina, and stable coronary disease), with atherosclerotic target lesion(s) in coronary arteries with visually estimated reference vessel diameters ≥2.25 mm and ≤4.0 mm.

DETAILED DESCRIPTION:
TARGET-IV NA trial is a prospective, multicenter, 1:1 randomized (Firehawk® vs. 2nd generation DES), trial.

Sub studies:

Angiographic sub study: The first approximately 200 consecutive consenting patients will be enrolled in the angiographic substudy. Optical coherence tomography (OCT) substudy: The first approximately 50 consecutive consenting subjects will be enrolled in the OCT substudy.

Clinical follow-up will be performed at 30 days, 6 months, and 1, 2, 3, 4, and 5 years post randomization. First approximately 200 consecutive consenting patients will undergo planned angiographic follow-up at 13 months after enrollment, with first 50 of these patients also consented to undergo planned OCT at baseline and at 13 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient understands the trial requirements and treatment procedures and provides written informed consent prior to any trial-specific tests or treatment.
3. Patients with an indication for PCI including angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or a positive coronary physiology test (e.g. FFR≤0.80 or iFR<0.90 or rFR ≤ 0.89 must be present), NSTEMI, or recent STEMI (STEMI >24 hours and in whom enzyme levels have peaked). For STEMI the time of presentation to the first treating hospital, whether a transfer facility or the study hospital, must be >24 hours prior to randomization and enzyme levels (CK-MB or Troponin) demonstrating that either or both enzyme levels have peaked.
4. Patient is willing to comply with all protocol-required follow-up evaluations.

Angiographic inclusion criteria:

1. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥2.25 mm to ≤4.0 mm and up to 44 mm in length.
2. The coronary anatomy is deemed likely to allow delivery of a study device to the target lesion(s).
3. Complex lesions are allowed including calcified lesions (lesion preparation is allowed and strongly recommended with current approved devices (e.g. scoring/cutting balloon and rotational/orbital atherectomy), multivessel disease, CTO,bifurcation lesions (except planned dual stent implantation), ostial lesions, tortuous lesions, and protected left main lesions.
4. Overlapping stents are allowed

Exclusion Criteria:

1. STEMI within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital or in whom enzyme levels (either CK-MB or Troponin) have not peaked.
2. PCI within the 24 hours preceding the baseline procedure.
3. History of stent thrombosis.
4. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
5. Subject is intubated.
6. Known LVEF <30%.
7. Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or the trial stent system or any protocol-required concomitant medications or devices (e.g. cobalt chromium alloy, stainless steel, sirolimus, everolimus or structurally related compounds, polymer, any P2Y12 inhibitor, or aspirin).
8. Planned surgery within 6 months.
9. Subject has an indication for chronic oral anticoagulant treatment (with either vitamin K antagonists or novel anticoagulants - NOACs)
10. Calculated creatinine clearance <30 mL/min using Cockcroft-Gault equation (<40 mL/min for subjects participating in the angiographic follow-up sub-study).
11. Hemoglobin <10 g/dL.
12. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
13. White blood cell (WBC) count <3,000 cells/mm3.
14. Clinically significant liver disease.
15. Active peptic ulcer or active bleeding from any site.
16. Other serious medical illness with a life-expectancy < 24 months (e.g. cancer, severe heart failure, severe lung disease).
17. A planned procedure that may cause non-compliance with the protocol or confound data interpretation.
18. Participation in another investigational drug or device trial that has not yet reached its primary endpoint and that may interfere with protocol compliance or confound data interpretation (as per the opinion of the investigator); or intent to participate in another investigational drug or device trial within 12 months.
19. Intention to become pregnant within 12 months (women of child-bearing potential who are sexually active must agree to use contraceptives from the time of enrollment through 12 months post-procedure).
20. Pregnancy or nursing (women of child-bearing potential must have a pregnancy test within 7 days prior to the index procedure).
21. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.).
22. Subject has received an organ transplant or is on a waiting list for an organ transplant.
23. Subject is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed.

Angiographic Exclusion Criteria:

1. Unprotected left main interventions
2. Bifurcation lesions with intended dual stent implantations
3. DES restenotic lesions
4. Prior PCI in the target vessel in the 12 months prior to enrollment
5. Any lesion in the target vessel that is likely to require PCI within 12 months
6. Stent lengths >36mm for diameters 2.0 mm and 2.25 mm (i.e., very long thin stents).
7. Lesion with intended ≥ 3 stent implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1720 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 months
  Percentage of participants that had either Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel)or Target Lesion Revascularization (TLR, clinically indicated) after one year

SECONDARY OUTCOMES:
In-stent late loss | 13 months
  In-stent late loss at 13 months post-procedure as measured by quantitative coronary angiography (QCA)
Neointimal thickness | 13 months
  Neointimal thickness at 3 months measured by Optical Coherence Tomography (OCT)
Target Lesion Failure | 12 months and yearly thereafter until 5 years
  Percentage of participants that had either Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel)or Target Lesion Revascularization (TLR, clinically indicated)
Target vessel failure | 12 months and yearly thereafter until 5 years
  Percentage of participants that had either cardiac death, target vessel-related MI*, or ischemia-driven target-vessel revascularization
Major adverse cardiac events (MACE) | 12 months and yearly thereafter until 5 years
  Percentage of participants that had either cardiac death, target vessel-related MI*, or ischemia-driven target-vessel revascularization
All-cause mortality | 12 months and yearly thereafter until 5 years
  mortality rate
Cardiac death | 12 months and yearly thereafter until 5 years
  Cardiac death rate
Q-wave MI | 12 months and yearly thereafter until 5 years
  percentage of participants that had Q-wave MI
Non Q-wave MI | 12 months and yearly thereafter until 5 years
  percentage of participants that had Non Q-wave MI
Any MI | 12 months and yearly thereafter until 5 years
  percentage of participants that had any MI
Target vessel MI | 12 months and yearly thereafter until 5 years
  percentage of participants that had MI related to target vessel
Any revascularization | 12 months and yearly thereafter until 5 years
  percentage of participants that had any revascularization
Ischemia-driven TLR | 12 months and yearly thereafter until 5 years
  percentage of participants that had Ischemia-driven TLR
Probable stent thrombosis | 12 months and yearly thereafter until 5 years
  percentage of participants that had Probable stent thrombosis
Definite stent thrombosis | 12 months and yearly thereafter until 5 years
  percentage of participants that had Definite stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Martin Leon, Study Chair — Columbia University
Locations (57):
- United States (44):
  - Cardiology PC, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - UC San Diego School of Medicine, La Jolla, California
  - Riverside Community Hospital, Riverside, California
  - Sharp Memorial Hospital, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Yale New Heaven Hospital, New Haven, Connecticut
  - JFK Medical Center, Atlantis, Florida
  - CCC Research - Countryside, Clearwater, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Atlanta Veterans Affairs Medical Center, Decatur, Georgia
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Eastern Maine Medical Center-Northern Light Cardiology, Bangor, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Inc., Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Bay, Bay City, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - McLaren Northern Michigan, Petoskey, Michigan
  - Metropolitan Heart Vascular Institute, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - St Dominic Hospital, Jackson, Mississippi
  - Boone Hospital Center, Columbia, Missouri
  - Bryan Medical Center East, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center/NYPH, New York, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Mercy Health St. Vincent Medical Center LLC, Toledo, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - UPMC Harrisburg Hospital, Harrisburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Texas Tech University Health, Lubbock, Texas
  - East Texas Medical Center, Tyler, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
  - Mayo Clinic Health System, La Crosse, Wisconsin
- Onze Lieve Vrouw Hospital, Aalst, Belgium
- Canada (7):
  - University of Calgary- Foothills Medical Center, Calgary, Alberta
  - St. Boniface Hospital Inc., Winnipeg, Manitoba
  - York PCI Group Inc, Newmarket, Ontario
  - IUPQ, Québec, Qebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - CIUSSE de l'estrie CHUS, Sherbrooke, Quebec
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Roskilde University Hospital, Roskilde
- Radbout UMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yeh RW, Bertrand OF, Mahmud E, Barbato E, Falah B, Issever MO, Redfors B, Popma A, Curtis M, van Royen N, Tanguay JF, Janssens L, Newman WN, Teeuwen K, Choi JW, Dirksen MT, Maehara A, Leon MB. Randomized Comparison of Novel Low-Dose Sirolimus-Eluting Biodegradable Polymer Stent vs Second-Generation DES: TARGET-IV NA Trial. J Am Coll Cardiol. 2025 Feb 18;85(6):563-574. doi: 10.1016/j.jacc.2024.10.074. Epub 2024 Oct 30. PMID 39480379